CLINICAL TRIAL: NCT04199052
Title: LinkPositively: A Technology-Delivered Peer Navigation and Social Networking Intervention to Improve HIV Care Across the Continuum for Black Women Affected by Interpersonal Violence
Brief Title: LinkPositively: A Technology-Delivered Peer Navigation and Social Networking Intervention to Improve HIV Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: San Diego State University (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Jamila K. Stockman, Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 191398; R34MH122014-01 (NIH)
Record Dates: First submitted 2019-12-09; First posted 2019-12-13 (Actual); Results first posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: HIV/AIDS
Keywords: HIV Care Continuum, Mobile Apps
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The investigators were blinded to participant study group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): Women assigned to the control arm will receive self-directed (non-Virtual Peer Navigator (PN) supported) treatment as usual at the HIV care service provider of choice following the Ryan White standard of care (i.e., referrals to physical, dental and mental health services; case management; and ancillary services. Annual assessments (e.g., updates on insurance, housing, referrals needed, behavioral assessment [e.g., depression, substance use]) are conducted by a case manager. For women who have fallen out of care and re-engage care, case management begins with an interview and assessment of current needs. Goals are set to create an individual care plan related to medical care, housing, and other resources, as needed. Referrals are made to appropriate services (e.g., primary care, housing, benefits counseling, food, support services) based on the intake assessment. It is important to note that the case management approach is self-guided versus intensive virtual PN assistance.
- LinkPositively Intervention (Experimental): Women assigned to the LinkPositively intervention arm will have access to all four components of the LinkPositively app. Women will be scheduled for a session with staff to inform them of their assigned virtual Peer Navigator (PN). Staff will train participants on how to download the app, explain the five components, using each component, and contacting their PN. Within the first week after, virtual PNs will complete a one-on-one, in-person or phone intake session with the participant, based on the participant's preference. During this intake session, the PN will conduct a participant needs assessment to connect her to HIV medical care via local health clinics and identify other areas of need, services of need, and assisted referrals (domestic violence services, mental health care, substance abuse treatment, housing and legal support, etc.). PNs will provide trauma-informed emotional and informational support, including guidance on accessing information about referred services.
  Interventions: Behavioral: LinkPositively

INTERVENTIONS:
Behavioral: LinkPositively — LinkPositively is a culturally tailored, trauma-informed smartphone app for Black women living with HIV/AIDS affected by interpersonal violence. Core components of LinkPositively include: a) Virtual Peer Navigation that includes phone and text check-ins and 4 weekly one-on-one video sessions to build skills to cope with barriers and navigate care; b) Social Networking platform to receive peer support; c) Educational and Self-care database with healthy living and self-care tips; d) GPS-enabled Resource Locator for HIV care and ancillary support service agencies; and e) ART self-monitoring and reminder system.
  Arms: LinkPositively Intervention

SUMMARY:
Investigators will develop and pilot test a culturally tailored, trauma-informed smartphone app, called LinkPositively, for Black WLHA affected by interpersonal violence. The goal is to determine preliminary effects of the intervention on HIV care (i.e., retention in HIV care, ART adherence) and mental health outcomes (e.g., PTSD, depression, anxiety). Through a randomized control trial (RCT), participants will be randomly assigned to either the intervention arm (n=40) or control arm (Ryan White standard of care, n=40), with follow-up at 3- and 6- months. This study will benefit the advancement of HIV prevention science by harnessing technology to promote engagement in HIV care, while improving social support through peers and social networking-all under the auspices of being trauma-informed for Black WLHA with experiences of interpersonal violence.

DETAILED DESCRIPTION:
In the US, Black women living with HIV/AIDS (WLHA) are less likely to be engaged in care, adherent to antiretroviral therapy (ART), and virally suppressed compared to White WLHA. Black women are also disproportionately affected by interpersonal violence - physical, sexual, and/or psychological abuse by a current or former intimate partner or non-intimate partner - which may co-occur with poor mental health and/or substance use, further contributing to ART non-adherence, lower CD4 counts, and reduced viral suppression. Peer Navigation, while highlighted as a successful model of care in improving HIV care outcomes, requires resources that HIV service agencies often lack. A scalable and sustainable solution is the use of mobile health (mHealth) smartphone applications ("apps"). Although there has been an increase in mHealth interventions developed for HIV prevention and care among at-risk and HIV-positive men who have sex with men (MSM) and youth, investigators are unaware of any to improve retention in care, ART adherence, and viral suppression among Black WLHA, nor any mHealth interventions that are responsive to Black women's experiences with interpersonal violence. To address this gap, investigators will develop and pilot test a culturally tailored, trauma-informed smartphone app, called LinkPositively, for Black WLHA affected by interpersonal violence. Core components of LinkPositively include: a) Virtual Peer Navigation that includes phone and text check-ins and 4 weekly one-on-one video sessions to build skills to cope with barriers and navigate care; b) Social Networking platform to receive peer support; c) Educational and Self-care database with healthy living and self-care tips; d) global positioning system-enabled Resource Locator for HIV care and ancillary support service agencies; and e) ART self-monitoring and reminder system. Guided by the Theory of Triadic Influences and Syndemic Theory, investigators will pilot test LinkPositively to assess preliminary effects of the intervention on HIV care (i.e., retention in care and ART adherence) and mental health outcomes (e.g., PTSD, depression, anxiety). Participants will be randomly assigned to either the intervention (n=40) or control (Ryan White standard of care, n=40) arm, with follow-up at 3- and 6- months. This study will benefit the advancement of HIV prevention science by harnessing technology to promote engagement in HIV care, while improving social support through peers and social networking - all under the auspices of being trauma-informed for Black WLHA with experiences of interpersonal violence.

ELIGIBILITY:
Inclusion Criteria:

* Female Gender
* Black or African-American racial/ethnic background
* Aged 18 years or older
* HIV-positive status
* Ever experienced physical, sexual, and/or psychological abuse by a current or former partner or non-partner (e.g., relative, friend, stranger)
* Owner of a smartphone with internet browsing capabilities
* English speaking

Exclusion Criteria:

* Male Gender
* Aged 17 or younger
* HIV-negative status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female gender identifying
Enrollment: 53 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jamila K. Stockman, PhD, MPH, Principal Investigator — University of California, San Diego; Keith J. Horvath, PhD, Principal Investigator — San Diego State University
Locations (1):
- UCSD AntiViral Research Center, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No
No current plan

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Although 53 participants were eligible and enrolled into the study, 10 elected not to participate following the informed consent process, resulting in a total of 43 participants continuing on in the study.
Groups:
- LinkPositively Intervention: Women assigned to the LinkPositively intervention arm will have access to all four components of the LinkPositively app. Core components of LinkPositively include: a) Virtual Peer Navigation that includes phone and text check-ins and 4 weekly one-on-one video sessions to build skills to cope with barriers and navigate care; b) Social Networking platform to receive peer support; c) Educational and Self-care database with healthy living and self-care tips; d) global positioning system-enabled Resource Locator for HIV care and ancillary support service agencies; and e) HIV medication self-monitoring and reminder system. Within the first week of the LinkPositively app use, virtual PNs will complete a one-on-one, in-person or phone intake session with the participant, based on the participant's preference. During this intake session, the PN will conduct a participant needs assessment to connect her to HIV medical care via local health clinics and identify other areas of need, services of need, and assisted referrals (domestic violence services, mental health care, substance abuse treatment, housing and legal support, etc.). Weekly, PNs will provide trauma-informed emotional and informational support, including guidance on accessing information about referred services.
Period: Overall Study
Arm/Group | Standard of Care | LinkPositively Intervention
Started | 17 | 26
Completed Intervention Period | 17 | 26
Completed 3-month Follow-up | 11 | 9
Completed | 6 | 8
Not Completed | 11 | 18
Not completed — Lost to Follow-up | 11 | 18

BASELINE CHARACTERISTICS:
Groups:
- LinkPositively Intervention: Women assigned to the LinkPositively intervention arm will have access to all four components of the LinkPositively app. Core components of LinkPositively include: a) Virtual Peer Navigation that includes phone and text check-ins and 4 weekly one-on-one video sessions to build skills to cope with barriers and navigate care; b) Social Networking platform to receive peer support; c) Educational and Self-care database with healthy living and self-care tips; d) GPS-enabled Resource Locator for HIV care and ancillary support service agencies; and e) ART self-monitoring and reminder system. Within the first week of LP app use, virtual PNs will complete a one-on-one, in-person or phone intake session with the participant, based on the participant's preference. During this intake session, the PN will conduct a participant needs assessment to connect her to HIV medical care via local health clinics and identify other areas of need, services of need, and assisted referrals (domestic violence services, mental health care, substance abuse treatment, housing and legal support, etc.). Weekly, PNs will provide trauma-informed emotional and informational support, including guidance on accessing information about referred services.
- Total: Total of all reporting groups
Arm/Group | Standard of Care | LinkPositively Intervention | Total
Number analyzed (Participants) | 17 | 26 | 43
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 49.50 [35.25 to 54.00] | 48.00 [33.50 to 55.25] | 49.00 [34.00 to 55.00]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 26 | 43
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 17 | 24 | 41
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 22 | 37
  White | 0 | 0 | 0
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17 | 26 | 43
Number of participants who have ever experienced physical violence [Count of Participants; unit: Participants] | 12 | 19 | 31
Number of participants who have ever experienced sexual assault [Count of Participants; unit: Participants] | 15 | 19 | 34
Number of participants who have ever experienced forced sexual activity [Count of Participants; unit: Participants] | 14 | 20 | 34
Number of participants who have ever experienced emotional abuse [Count of Participants; unit: Participants] | 17 | 25 | 42
Number of participants who have ever experienced attempts to control you [Count of Participants; unit: Participants] | 13 | 22 | 35
Number of participants who have experienced threats of physical violence [Count of Participants; unit: Participants] | 13 | 18 | 31
Number of HIV Care Visits in Past Year [Median (Inter-Quartile Range); unit: HIV care visits] | 3.00 [2.00 to 4.50] | 2 [2.00 to 4.00] | 2.00 [2.00 to 4.00]
HIV Adherence Self-Efficacy [Median (Inter-Quartile Range); unit: units on a scale] — HIV Adherence Self-Efficacy measured using the HIV Adherence Self-Efficacy Scale, minimum=0, maximum=10; higher scores mean greater self-efficacy to adhere to HIV medication.
  units on a scale | 8.67 [5.17 to 9.67] | 8.17 [6.45 to 9.69] | 8.25 [6.33 to 9.67]
National Stress Events Survey PTSD Short Scale [Median (Inter-Quartile Range); unit: units on a scale] — PTSD is measured using the National Stressful Events Survey PTSD Short Scale, minimum value=0, maximum value=36; higher scores indicate a worse outcome (greater PTSD symptomatology).
  units on a scale | 13.00 [6.00 to 19.50] | 10.00 [7.00 to 19.00] | 11.00 [7.00 to 19.00]
Patient Health Questionnaire for Depression [Median (Inter-Quartile Range); unit: units on a scale] — Patient Health Questionnaire (PHQ-9) for depression symptoms. Score range minimum = 0, maximum = 27, with higher scores indicating more depressive symptoms
  units on a scale | 9.00 [6.00 to 12.00] | 9.00 [4.00 to 12.25] | 9.00 [6.00 to 12.00]
Generalized Anxiety Disorder [Median (Inter-Quartile Range); unit: units on a scale] — Generalized Anxiety Disorder (GAD-7) for anxiety symptoms. Score ranges from minimum = 0, maximum = 21, with higher scores indicating more anxiety symptoms
  units on a scale | 7.00 [5.00 to 11.50] | 7.00 [5.50 to 12.50] | 7.00 [5.00 to 12.00]

OUTCOME MEASURES:

1. Primary Outcome: Number of HIV Care Visits
Description: Median number of HIV care visits
Time Frame: 3 Months Post-Baseline
Measure: Median (Inter-Quartile Range); unit: HIV Care Visits
Arm/Group | Standard of Care | LinkPositively Intervention
Number analyzed (Participants) | 11 | 9
HIV Care Visits | 1.00 [1.00 to 2.00] | 3.00 [0.50 to 3.00]

2. Primary Outcome: Number of HIV Care Visits
Description: Median number of HIV care visits in past 6 months
Time Frame: 6 Months Post-Baseline
Measure: Median (Inter-Quartile Range); unit: HIV Care Visits
Arm/Group | Standard of Care | LinkPositively Intervention
Number analyzed (Participants) | 6 | 8
HIV Care Visits | 2.00 [1.00 to 3.50] | 3.00 [1.00 to 5.00]

3. Primary Outcome: Number of Participants With ART Adherence
Description: Dichotomized into two groups (Greater than or equal to 90% adherence to ART regime (self-report) based on the Wilson 3-item adherence self-report items vs. Less than 90% adherence to ART regime (self-report) based on the Wilson 3-item adherence self-report items)
Time Frame: 3 Months Post-Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | LinkPositively Intervention
Number analyzed (Participants) | 11 | 9
Participants | 8 | 7

4. Primary Outcome: Number of Participants With ART Adherence
Description: as for outcome 3
Time Frame: 6 Months Post-Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | LinkPositively Intervention
Number analyzed (Participants) | 6 | 8
Participants | 3 | 7

5. Primary Outcome: HIV Adherence Self-Efficacy
Description: HIV Adherence Self-Efficacy measured using the HIV Adherence Self-Efficacy Scale, minimum=0, maximum=10; higher scores mean greater self-efficacy to adhere to HIV medication.
Time Frame: 3 Months Post-Baseline
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Standard of Care | LinkPositively Intervention
Number analyzed (Participants) | 11 | 9
units on a scale | 8.17 [6.58 to 9.67] | 8.33 [6.96 to 9.79]

6. Primary Outcome: HIV Adherence Self-Efficacy
Description: as for outcome 5
Time Frame: 6 Months Post-Baseline
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Standard of Care | LinkPositively Intervention
Number analyzed (Participants) | 6 | 8
score on a scale | 8.21 [6.79 to 9.31] | 9.18 [6.79 to 9.42]

7. Secondary Outcome: National Stressful Events Survey PTSD Short Scale Score
Description: PTSD is measured using the National Stressful Events Survey PTSD Short Scale, minimum value=0, maximum value=36; higher scores indicate a worse outcome (greater PTSD symptomatology).
Time Frame: 3 Months Post-Baseline
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Standard of Care | LinkPositively Intervention
Number analyzed (Participants) | 11 | 9
score on a scale | 12.00 [2.00 to 20.00] | 8.00 [5.50 to 16.50]

8. Secondary Outcome: National Stressful Events Survey PTSD Short Scale Score
Description: as for outcome 7
Time Frame: 6 Months Post-Baseline
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Standard of Care | LinkPositively Intervention
Number analyzed (Participants) | 6 | 8
score on a scale | 10.00 [3.75 to 18.75] | 7.50 [5.25 to 12.75]

9. Secondary Outcome: Patient Health Questionnaire for Depression Score
Description: Measured using the Patient Health Questionnaire-9, minimum value=0, maximum value=27; higher scores indicate more depression.
Time Frame: 3 Months Post-Baseline
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Standard of Care | LinkPositively Intervention
Number analyzed (Participants) | 11 | 9
score on a scale | 7.00 [4.00 to 12.00] | 6.00 [4.00 to 7.50]

10. Secondary Outcome: Patient Health Questionnaire for Depression Score
Description: Measured using Patient Health Questionnaire-9, minimum value=0, maximum value=27; higher scores indicate more depression.
Time Frame: 6 Months Post-Baseline
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Standard of Care | LinkPositively Intervention
Number analyzed (Participants) | 17 | 26
score on a scale | 8.50 [6.75 to 11.25] | 6.00 [1.50 to 8.75]

11. Secondary Outcome: Generalized Anxiety Disorder Score
Description: Anxiety measured using the Generalized Anxiety Disorder Scale-7, minimum value=0, maximum value=21; higher scores mean a worse outcome.
Time Frame: 3 Months Post-Baseline
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Standard of Care | LinkPositively Intervention
Number analyzed (Participants) | 11 | 9
score on a scale | 6.00 [2.00 to 11.00] | 6.00 [4.50 to 8.00]

12. Secondary Outcome: Generalized Anxiety Disorder Score
Description: Anxiety was measured using the Generalized Anxiety Disorder Scale-7, minimum value=0, maximum value=21; higher scores mean a worse outcome.
Time Frame: 6 Months Post-Baseline
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Standard of Care | LinkPositively Intervention
Number analyzed (Participants) | 6 | 8
score on a scale | 8.00 [2.75 to 11.00] | 5.00 [3.25 to 7.75]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over a 6 month period.
Arm/Group | Standard of Care | LinkPositively Intervention
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/26
Other Adverse Events (participants affected / at risk) | 0/17 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-05-01): https://cdn.clinicaltrials.gov/large-docs/52/NCT04199052/Prot_SAP_000.pdf